CLINICAL TRIAL: NCT05740384
Title: Assessing the Sensitivity and Specificity of Sonotubometry to Measure the Eustachian Tube Function
Brief Title: The Accuracy of Sonotubometry to Assess the Eustachian Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: James Tysome (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor-Investigator, James Tysome, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A096497
Record Dates: First submitted 2023-01-31; First posted 2023-02-23 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Eustachian Tube Dysfunction
Keywords: obstructive Eustachian tube dysfunction; Eustachian tube dysfunction

STUDY DESIGN:
Intervention Model Description: This is a validation study in 28 ears with Eustachian tube dysfunction.
Masking Description: The order of the assessment measurements is batch-wise randomised but there is no masking. Both the participant and investigator know what sort of measurements is being performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sonotubometry Assessment (Experimental): All participants will be measured 8 times using sonotubometry. 2 times without applying any sound and 2 times while applying sound. This is done for both the left and right ear.
  Interventions: Device: Sonotubometry Assessment

INTERVENTIONS:
Device: Sonotubometry Assessment — The exact order of the measurements will be randomised:
  * Recording type 1: No sound applied, 10 seconds recording of baseline noise, followed by recording when the participant is asked to swallow 3 times.
  * Recording type 2: White noise applied, 10 seconds recording of baseline noise, followed by recording when the participant is asked to swallow 3 times.
  * Ask for subjective feedback (did you hear a change in the sound in your ear on swallowing?) after each recording
  * This is repeated using the contralateral ear and nostril. After successful recording, the microphone will be removed.
  For comparison, tubomanometry measurements will be performed on each ear. Tubomanometry is an alternative method to assess the middle ear and Eustachian tube. Afterwards, the participant's involvement in the study will be complete. The entire involvement will take about 50 minutes.

SUMMARY:
The Eustachian tube (ET) connects the middle ear with the throat and is important for maintaining a healthy middle ear. Sonotubometry is a new method to measure how well the ET works by using sound. A speaker is placed at the nostril and a microphone records sound in the external ear canal. The ET is closed at rest and opens with swallowing. This is measured as an increase in sound measured in the external ear by sonotubometry.

Previous research has not proven that sonotubometry is reliable enough to be used in clinics to assess ET dysfunction (a disease where the ET does not open properly). In a recent study with healthy volunteers, it was possible to identify many of the existing issues of sonotubometry and improve the reliability of this method. This was primarily achieved by testing different sound types and sound volumes. This study aims to assess the reliability and usability of the new testing protocol in study participants with ET dysfunction. The results of this study will then be compared with the results from the previous study with healthy volunteers to work out how well sonotubometry works. Ultimately, this research aims to improve the ability to diagnose ET dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Participant is capable of giving informed consent (in the English language)
* Participant has a current diagnosis of obstructive Eustachian tube dysfunction in the ear clinic at Addenbrooke's Hospital
* Age 16 and over

Exclusion Criteria:

* Cardiac pacemaker (incompatible with the large sonotubometry speaker magnet)
* Discharging or infected ear (for infection control reasons)
* Otitis Media with effusion (complicates test interpretation)
* Cleft palate or Craniofacial abnormalities (complicates test interpretation)
* Cholesteatoma (complicates test interpretation)
* Nasopharyngeal mass (complicates test interpretation)
* History of radiotherapy to the head and neck (can affect surrounding tissue structure)

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Assess Specificity and Sensitivity of Sonotubometry using a Custom-Built Sonotubometer | 40-50 minutes
  The main objective of the trial is to measure the specificity and sensitivity of an assessment method of the Eustachian tube called sonotubometry. To do this, eight sonotubometry measurements will be performed on each patient using the custom built Sonotubometry device. In total a maximum of 28 patients will be measured. This data will be compared to measurements from volunteers (data collected through a different study) to measure the sensitivity and specificity in percentage.

SECONDARY OUTCOMES:
Ability of Sonotubometry Measurements to detect Eustachian tube opening by using an Increased Sound Amplitude | 40-50 minutes
  The secondary objective is to assess if sonotubometry with an sound amplitude of 120dB is able to detect Eustachian tube opening. In the past a lower sound level was used (below 110dB) and thus the goal here is to measure the suitability of a higher sound pressure for sonotubometry. This will be measured by the ability of the new method to reliably detect the Eustachian tube function in patients and healthy volunteers (healthy volunteers data was gathered in a separate study)

CONTACTS AND LOCATIONS:
Overall Officials: James Tysome, Dr, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided